CLINICAL TRIAL: NCT07237451
Title: Cardiovascular and Renal Endpoints With Flozins - an Observational Prospective Study in CKD HFpEF Patients
Acronym: CARE FOR CKD H
Status: Recruiting | Type: Observational
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: Dr. C.I. Parhon Hospital, Iasi (Unknown); The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Adrian Covic, Professor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: CARE FOR CKD HFPEF
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: CKD - Chronic Kidney Disease; Heart Failure Preserved Ejection Fraction; SGLT2 Inhibitors; Diabetes (DM)
Keywords: CKD; HFpEF; SGTL2 inhibitors; Biomarkers; PWV
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure, Diastolic; Diabetes Mellitus | interventions — Vascular Stiffness; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iSGLT2 therapy: CKD and HFpEF with iSGLT2 therapy
  Interventions: Diagnostic Test: Arterial stiffness; Diagnostic Test: Echocardiography; Other: Biomarkers determination; Other: NMR metabolomics and uremic toxins mapping
- Control: CKD and HFpEF without iSGLT2 therapy
  Interventions: Diagnostic Test: Arterial stiffness; Diagnostic Test: Echocardiography; Other: Biomarkers determination; Other: NMR metabolomics and uremic toxins mapping

INTERVENTIONS:
Diagnostic Test: Arterial stiffness — Arterial stiffness assessment will be performed by applanation tonometry with the patient being recumbent, 10 minutes before the measures were done. The carotid and femoral pulse will be acquired by applanation tonometry sequentially, allowing a single operator to acquire the measurement. The transit time from the R-wave of the simultaneously acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference between these 2 transit times is divided by distances measured from the body surface to estimate the arterial path length in order to calculate carotid-femoral PWV.
Diagnostic Test: Echocardiography — Echocardiography will be performed on each patient at baseline; the measurements will be carried out according to the recommendations of the American Society of Echocardiography. Echocardiographic evaluation will provide information about cardiac anatomy (e.g. volumes, geometry, mass) and function (e.g. left ventricular function and wall motion, valvular function, right ventricular function, pulmonary artery pressure, pericardium).
Other: Biomarkers determination — NT-pro BNP, Syndecan-1, VCAM-1, Endoglin, NO and ADMA will be determined by specific enzyme linked immunosorbent assay (ELISA) kits.
Other: NMR metabolomics and uremic toxins mapping — The aliquoted serum preserved at -80° C will be analysed by NMR using deuterated solvents (D2O, CDCl3, CD3OD, CD3CN), standards of metabolites and uremic toxins.

SUMMARY:
The main aim of this study is to holistically assess the cardiovascular and renal outcomes in HFpEF CKD patients with and without SGLT2 inhibition, with focus on the endothelial disfunction, MACE and mortality using clinical evaluation, flow mediated dilatation, carotid-femoral pulse wave velocity, intima-media thickness, echocardiographic parameters, NMR metabolomics and a series of novel biomarkers.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is considered to become the 5th cause of death worldwide by 2040. Aging populations, growing frequency of type 2 diabetes, hypertension, a low detection rate and therapeutic inertia in the early stages of CKD determined the increasing incidence and prevalence. CKD patients exhibit an elevated cardiovascular risk manifesting myocardial infarction and stroke, coronary artery disease, heart failure (HF), arrhythmias, and sudden cardiac death. The relationship between HF and CKD is bidirectional, with chronic HF promoting CKD development (cardio-renal syndrome type 1), and CKD promoting the development of HF (type 3). In the last decade, HF with preserved ejection fraction (HFpEF) represents the typical phenotype in patients with CKD, accounting for more than half of the cases of HF. Given the high burden of both HF and CKD, their complex interaction and challenging management, along with the prognostic implications regarding comorbidity and mortality, a comprehensive approach in the HFpEF population is mandatory, since HF diagnosis was evasive for years. The main aim of this study is to holistically assess the cardiovascular and renal outcomes in HFpEF CKD patients with and without SGLT2 inhibition, with focus on the endothelial disfunction, MACE and mortality using clinical evaluation, flow mediated dilatation, carotid-femoral pulse wave velocity, intima-media thickness, echocardiographic parameters, NMR metabolomics and a series of novel biomarkers.

The objectives of this prospective observational study are to determine:

* the feasibility of PWV measurement and ventricular strain in HFpEF CKD patients with and without SGLT2 inhibition;
* the cardiovascular outcomes, namely MACE, defined as time to first non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure or CV death and on all-cause mortality in HFpEF CKD patients with and without SGLT2 inhibition;
* the renal outcomes, such as rapid progression of renal disease - defined as sustained annual decline of at least 5mL/min/1,73m2 in eGFR or a sustained drop of 25% or more in eGFR within 12 months;
* the metabolomics profile related to uremic toxins panel determined by NMR spectroscopy and other biological markers as novel molecules with a higher potential accuracy of predicting further major cardiovascular events in HFpEF CKD patients with and without SGLT2 inhibition.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years;
* ejection fraction > 40;
* patients with CKD stage 3-4 (eGFR between 15-60 mL/min/1.73m2), with iSGLT2 recommendation, diabetic and non-diabetic;
* age, sex and CKD stage 3 and 4 matched patients without iSGLT2 administration.

Exclusion Criteria:

* eGFR< 15 mL/min/1.73m2 or patients undergoing dialysis;
* presence of congenital heart disease, decompensated cirrhosis, pregnancy and active malignancies;
* coronary artery disease (including those with a history of acute coronary syndrome, angina pectoris, or prior coronary angiography or CT angiography demonstrating significant coronary artery lesions);
* cardiac medical devices, namely metallic joint prostheses, cardiac stent or pacemakers;
* active systemic infections (due to interference with biomarkers that can give false rise values).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD stages 3 and 4 (eGFR calculated by CKD-EPI) with HFpEF
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 20 months
  Composite CV outcome: time to first non-fatal myocardial infarction, non-fatal stroke, and hospitalization for heart failure or CV death
All-cause mortality | 10 and 20 months
  All-cause mortality

SECONDARY OUTCOMES:
Composite renal outcome | 10 and 20 months
  Rapid progression of renal disease - defined as sustained annual decline of at least 5mL/min/1,73m2 in eGFR or a sustained drop of 25% or more in eGFR within 10 months

OTHER OUTCOMES:
Changes in cardiac biomarkers | Baseline, 10 and 20 months
  Blood levels of NT-pro BNP, Syndecan-1, VCAM-1, Endoglin, NO and ADMA will be measured at baseline and months 10 and 20. The outcome is defined as the change from baseline.
Changes in the NMR metabolomics and uremic toxins mapping | Baseline, 10 and 20 months
  Blood levels of NMR metabolomics and uremic toxins will be measured at baseline and months 10 and 20. The outcome is defined as the change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. C.I. Parhon Hospital in Iasi, Iași, Romania

IPD SHARING:
Plan to Share IPD: Undecided